CLINICAL TRIAL: NCT06249932
Title: The Safety and Efficacy of Empagliflozin in Patients with End-stage Renal Disease and Heart Failure with Reduced Ejection Fraction - a Randomized Controlled Trial
Brief Title: Empagliflozin in Heart Failure with Reduced Ejection Fraction and End Stage Renal Disease
Acronym: EMPA-RRED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202301140MINC
Record Dates: First submitted 2024-01-19; First posted 2024-02-08 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure with Reduced Ejection Fraction; End Stage Renal Disease on Dialysis
Keywords: end stage renal disease; sodium-glucose co-transporter 2 inhibitors,; heart failure with reduced ejection fraction; empagliflozin; left ventricular mass
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- empagliflozin (Experimental): Jardiance, 25 mg, QD, for 6 months
  Interventions: Drug: Empagliflozin 25 MG
- placebo (Placebo Comparator): QD, for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — The medication will be packed in a customized sealed jar and labeled on the exterior of the jar.
  Other Names: Jardiance® 25mg Film-Coated Tablets
  Arms: empagliflozin
Drug: Placebo — The placebo tablet is manufactured by Prince Pharmaceutical Co., Ltd, a leading manufacturer of nutritional supplements with certifications including cGMP, GMP, ISO, and HACCP. The Prince Pharmaceutical also provides Original Equipment Manufacturing (OEM)/Original Design Manufacturing (ODM) services for a wide array of tablet shapes, and post-processing techniques such as film coating and sugar coating.
  Arms: placebo

SUMMARY:
In patients with ESRD, up to 20% of patients suffer from HFrEF, leading to significant CV morbidity and mortality. Several drug classes that provide survival benefits for patients with HFrEF, including SGLT2i, lack data regarding their efficacy and safety in patients under chronic hemodialysis. As the primary target of SGLT2i is expressed mostly in the kidneys, the efficacy of SGLT2i in patients with ESRD may be limited. On the other hand, patients with ESRD are at higher risks of experiencing cardiovascular events and may still benefit from treatment. Several mechanistic studies have demonstrated direct actions of SGLT2i on the myocardium, thus it is possible that the benefits of SGLT2i on heart failure are independent of their glycosuric actions and may still be present in anuric subjects. Furthermore, pharmacokinetics and pharmacodynamics studies on empagliflozin demonstrated that peak plasma levels of empagliflozin in subjects with renal failure/ESRD were similar to those in subjects with normal renal function. The use of empagliflozin in patients with ESRD seemed safe in terms of pharmacokinetics and pharmacodynamics, yet its efficacy remains to be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years old
* ESRD under chronic, maintenance hemodialysis with stable dry weight for the past 6 months
* Documented left ventricular ejection fraction <50% by any imaging modality within 1 month of screening

Exclusion Criteria:

* Age <20 years old
* Ongoing pregnancy
* NYHA class IV heart failure
* Any hospitalization for heart failure within the past month
* Ongoing acute urinary tract infection at the time of screening
* Known acute genital infection
* Severe peripheral artery disease (Rutherford category 4-6)
* Acute coronary syndrome, stroke or transient ischemic attack within the past month
* Recent initiation of chronic maintenance hemodialysis within 6 months
* Adjustment of dry weight with changes greater than 5% of body weight within the past month
* Documented left ventricular ejection fraction ≥50% by any imaging modality within 1 month of screening
* Refused informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass | 24 weeks of treatment
  As assessed by cardiac magnetic resonance imaging, performed on non-dialysis day

SECONDARY OUTCOMES:
Left ventricular mass index | 24 weeks of treatment
  As assessed by cardiac magnetic resonance imaging, performed on non-dialysis day
LV end-systolic volume index | 24 weeks of treatment
  As assessed by cardiac magnetic resonance imaging, performed on non-dialysis day
LV end-diastolic volume index | 24 weeks of treatment
  As assessed by cardiac magnetic resonance imaging, performed on non-dialysis day
LA volume index | 24 weeks of treatment
  As assessed by cardiac magnetic resonance imaging, performed on non-dialysis day
LV ejection fraction | 24 weeks of treatment
  As assessed by cardiac magnetic resonance imaging, performed on non-dialysis day
Global longitudinal strain | 24 weeks of treatment
  As assessed by cardiac magnetic resonance imaging, performed on non-dialysis day
LV end-systolic volume index | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
LV end-diastolic volume index | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
LA volume index | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
LV ejection fraction | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Left ventricular mass index | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Global longitudinal strain | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
LV relative wall thickness | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Mitral early (E) and late (A) diastolic filling velocity ratio (E/A) | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Mitral inflow deceleration time | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
Tricuspid regurgitation peak gradient (TRPG) | 12 weeks and 24 weeks of treatment
  As assessed by echocardiography, performed on non-dialysis day
NT-proBNP | 4 weeks, 12 weeks and 24 weeks of treatment
  Blood tests obtained pre-dialysis session
HbA1c | 4 weeks, 12 weeks and 24 weeks of treatment
  Blood tests obtained pre-dialysis session
Lipid profile | 4 weeks, 12 weeks and 24 weeks of treatment
  Blood tests obtained pre-dialysis session
KCCQ-OS | 12 weeks and 24 weeks of treatment
  Performed on non-dialysis day
6-minute walking distance | 12 weeks and 24 weeks of treatment
  Performed on non-dialysis day
3-minute heart rate variability | 12 weeks and 24 weeks of treatment
  During hemodialysis session
Blood pressure | 12 weeks and 24 weeks of treatment
  Obtained pre-dialysis session
Major adverse cardiovascular events (composite of CV death, myocardial infarction, stroke) | 24 weeks of treatment
  By medical record confirmation and by interview
Lower extremity non-traumatic amputation or revascularization | 24 weeks of treatment
  By medical record confirmation and by interview
All-cause mortality | 24 weeks of treatment
  By medical record confirmation and by interview
Hospitalization for heart failure | 24 weeks of treatment
  By medical record confirmation and by interview
Hypoglycemic events | 24 weeks of treatment
  By medical record confirmation and by interview
Hypokalemia | 4 weeks, 12 weeks and 24 weeks of treatment
  Blood tests obtained pre-dialysis session
Diabetic ketoacidosis | 24 weeks of treatment
  By medical record confirmation and by interview
Urinary tract infection | 24 weeks of treatment
  By medical record confirmation and by interview
Genital tract infection | 24 weeks of treatment
  By medical record confirmation and by interview

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shu-Han Lin, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital; Chih-Cheng Wu, MD. PhD, Principal Investigator — National Taiwan University Hsin-Chu Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital Hsinchu Branch, Hsinchu, Taiwan
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ronco C, Haapio M, House AA, Anavekar N, Bellomo R. Cardiorenal syndrome. J Am Coll Cardiol. 2008 Nov 4;52(19):1527-39. doi: 10.1016/j.jacc.2008.07.051. PMID 19007588
- [Background] Bansal N, Zelnick L, Bhat Z, Dobre M, He J, Lash J, Jaar B, Mehta R, Raj D, Rincon-Choles H, Saunders M, Schrauben S, Weir M, Wright J, Go AS; CRIC Study Investigators. Burden and Outcomes of Heart Failure Hospitalizations in Adults With Chronic Kidney Disease. J Am Coll Cardiol. 2019 Jun 4;73(21):2691-2700. doi: 10.1016/j.jacc.2019.02.071. PMID 31146814
- [Background] Kotecha D, Gill SK, Flather MD, Holmes J, Packer M, Rosano G, Bohm M, McMurray JJV, Wikstrand J, Anker SD, van Veldhuisen DJ, Manzano L, von Lueder TG, Rigby AS, Andersson B, Kjekshus J, Wedel H, Ruschitzka F, Cleland JGF, Damman K, Redon J, Coats AJS; Beta-Blockers in Heart Failure Collaborative Group. Impact of Renal Impairment on Beta-Blocker Efficacy in Patients With Heart Failure. J Am Coll Cardiol. 2019 Dec 10;74(23):2893-2904. doi: 10.1016/j.jacc.2019.09.059. PMID 31806133
- [Background] Ferro CJ, Mark PB, Kanbay M, Sarafidis P, Heine GH, Rossignol P, Massy ZA, Mallamaci F, Valdivielso JM, Malyszko J, Verhaar MC, Ekart R, Vanholder R, London G, Ortiz A, Zoccali C. Lipid management in patients with chronic kidney disease. Nat Rev Nephrol. 2018 Dec;14(12):727-749. doi: 10.1038/s41581-018-0072-9. PMID 30361677
- [Background] Roehm B, Gulati G, Weiner DE. Heart failure management in dialysis patients: Many treatment options with no clear evidence. Semin Dial. 2020 May;33(3):198-208. doi: 10.1111/sdi.12878. Epub 2020 Apr 13. PMID 32282987
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Verma S, Mazer CD, Yan AT, Mason T, Garg V, Teoh H, Zuo F, Quan A, Farkouh ME, Fitchett DH, Goodman SG, Goldenberg RM, Al-Omran M, Gilbert RE, Bhatt DL, Leiter LA, Juni P, Zinman B, Connelly KA. Effect of Empagliflozin on Left Ventricular Mass in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease: The EMPA-HEART CardioLink-6 Randomized Clinical Trial. Circulation. 2019 Nov 19;140(21):1693-1702. doi: 10.1161/CIRCULATIONAHA.119.042375. Epub 2019 Aug 22. PMID 31434508
- [Background] Ersboll M, Jurgens M, Hasbak P, Kjaer A, Wolsk E, Zerahn B, Brandt-Jacobsen NH, Gaede P, Rossing P, Faber J, Inzucchi SE, Gustafsson F, Schou M, Kistorp C. Effect of empagliflozin on myocardial structure and function in patients with type 2 diabetes at high cardiovascular risk: the SIMPLE randomized clinical trial. Int J Cardiovasc Imaging. 2022 Mar;38(3):579-587. doi: 10.1007/s10554-021-02443-5. Epub 2021 Oct 20. PMID 34669059
- [Background] Soga F, Tanaka H, Tatsumi K, Mochizuki Y, Sano H, Toki H, Matsumoto K, Shite J, Takaoka H, Doi T, Hirata KI. Impact of dapagliflozin on left ventricular diastolic function of patients with type 2 diabetic mellitus with chronic heart failure. Cardiovasc Diabetol. 2018 Oct 8;17(1):132. doi: 10.1186/s12933-018-0775-z. PMID 30296931
- [Background] Li X, Lu Q, Qiu Y, do Carmo JM, Wang Z, da Silva AA, Mouton A, Omoto ACM, Hall ME, Li J, Hall JE. Direct Cardiac Actions of the Sodium Glucose Co-Transporter 2 Inhibitor Empagliflozin Improve Myocardial Oxidative Phosphorylation and Attenuate Pressure-Overload Heart Failure. J Am Heart Assoc. 2021 Mar 16;10(6):e018298. doi: 10.1161/JAHA.120.018298. Epub 2021 Mar 13. PMID 33719499
- [Background] Pabel S, Wagner S, Bollenberg H, Bengel P, Kovacs A, Schach C, Tirilomis P, Mustroph J, Renner A, Gummert J, Fischer T, Van Linthout S, Tschope C, Streckfuss-Bomeke K, Hasenfuss G, Maier LS, Hamdani N, Sossalla S. Empagliflozin directly improves diastolic function in human heart failure. Eur J Heart Fail. 2018 Dec;20(12):1690-1700. doi: 10.1002/ejhf.1328. Epub 2018 Oct 17. PMID 30328645
- [Background] Macha S, Mattheus M, Halabi A, Pinnetti S, Woerle HJ, Broedl UC. Pharmacokinetics, pharmacodynamics and safety of empagliflozin, a sodium glucose cotransporter 2 (SGLT2) inhibitor, in subjects with renal impairment. Diabetes Obes Metab. 2014 Mar;16(3):215-22. doi: 10.1111/dom.12182. Epub 2013 Aug 19. PMID 23859488
- [Background] He Z, Lam K, Zhao W, Yang S, Li Y, Mo J, Gao S, Liang D, Qiu K, Huang M, Wu J. SGLT-2 inhibitors and euglycemic diabetic ketoacidosis/diabetic ketoacidosis in FAERS: a pharmacovigilance assessment. Acta Diabetol. 2023 Mar;60(3):401-411. doi: 10.1007/s00592-022-02015-6. Epub 2022 Dec 28. PMID 36576563
- [Background] Jurgens M, Schou M, Hasbak P, Kjaer A, Wolsk E, Zerahn B, Wiberg M, Brandt NH, Gaede PH, Rossing P, Faber J, Inzucchi S, Gustafsson F, Kistorp CM. Design of a randomised controlled trial of the effects of empagliflozin on myocardial perfusion, function and metabolism in type 2 diabetes patients at high cardiovascular risk (the SIMPLE trial). BMJ Open. 2019 Nov 27;9(11):e029098. doi: 10.1136/bmjopen-2019-029098. PMID 31780586
- [Derived] Lin DS, Lo HY, Yang CW, Wu CC. Safety and Short-Term Effects of Empagliflozin in Patients with Heart Failure and End-Stage Renal Disease. Am J Cardiovasc Drugs. 2025 Aug 25. doi: 10.1007/s40256-025-00760-x. Online ahead of print. PMID 40855136